CLINICAL TRIAL: NCT02773368
Title: A Clinical Trial Comparing Glycaemic Control and Safety of Insulin Degludec/Liraglutide (IDegLira) Versus Insulin Glargine (IGlar) as add-on Therapy to SGLT2i in Subjects With Type 2 Diabetes Mellitus. DUALTM IX - Add-on to SGLT2i
Brief Title: A Clinical Trial Comparing Glycaemic Control and Safety of Insulin Degludec/Liraglutide (IDegLira) Versus Insulin Glargine (IGlar) as add-on Therapy to SGLT2i in Subjects With Type 2 Diabetes Mellitus
Acronym: DUALTM IX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4229; 2015-001596-48 (EudraCT Number); U1111-1168-9343 (Other: WHO); REec-2016-2248 (Other: REec)
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegLira (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- IGlar (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/liraglutide — IDegLira will be given subcutaneously ( s.c., under the skin) once daily.
  Arms: IDegLira
Drug: insulin glargine — IGlar will be given subcutaneously ( s.c., under the skin) once daily.
  Arms: IGlar

SUMMARY:
This trial is conducted globally. The aim of this trial is comparing glycaemic control and safety of insulin degludec/liraglutide (IDegLira) versus insulin glargine (IGlar) as add-on therapy to SGLT2i (sodium-glucose cotransporter 2 inhibitors) in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age at least 18 years at the time of signing informed consent - Subjects diagnosed (clinically) with type 2 diabetes mellitus - HbA1c 7.0-11.0% [53-97 mmol/mol] (both inclusive) by central laboratory analysis - Body mass index (BMI) equal to or above 20 kg/m^2 and below 40 kg/m^2 - Insulin naïve subjects; however short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as well as prior insulin treatment for gestational diabetes - A stable daily dose for at least 90 days prior to the day of screening of any SGLT2i in monotherapy or in combination with metformin ± DPP4i ± pioglitazone. Use of pioglitazone is not allowed in subjects treated with dapagliflozin Exclusion Criteria: - Receipt of any investigational medicinal product within 90 days prior to screening - Use of any OADs (other than SGLT2i in monotherapy or in combination with metformin or DPP4i or pioglitazone as described in the inclusion criteria) within 90 days prior to the day of screening - Use of glucagon-like peptide-1 (GLP-1) receptor agonist (e.g., exenatide or liraglutide) within 90 days prior to the day of screening - Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent severe metabolic dysregulation (e.g., diabetes ketoacidosis) in the previous 90 days prior to the day of the screening - Subjects presently classified as being in NYHA (New York Heart Association) Class III or IV1 - Renal impairment estimated Glomerular Filtration Rate 60 mL/min/1.73 m2 as per CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) - Impaired liver function, defined as ALT (alanine aminotransferase) equal to or above 2.5 times upper normal limit at screening - Known or suspected hypersensitivity to trial product(s) or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (83):
- United States (24):
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Mission Viejo, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Chiefland, Florida
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Bristol, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Mendoza
- Canada (6):
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Rovaniemi
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- Hungary (6):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Komárom
  - Novo Nordisk Investigational Site, Salgótarján
  - Novo Nordisk Investigational Site, Szekszárd
  - Novo Nordisk Investigational Site, Zalaegerszeg
- India (9):
  - Novo Nordisk Investigational Site, Hyderbad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bhopal, Madhya Pradesh
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Varanasi, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Russia (5):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Petesburg
- Slovakia (5):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Nitra
  - Novo Nordisk Investigational Site, Prešov
  - Novo Nordisk Investigational Site, Trnava
- Slovenia (5):
  - Novo Nordisk Investigational Site, Celje
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Kranj
  - Novo Nordisk Investigational Site, Murska Sobota
  - Novo Nordisk Investigational Site, Trbovlje
- Spain (6):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Boadilla del Monte
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Villamartín
- Switzerland (8):
  - Novo Nordisk Investigational Site, Baden
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lucerne
  - Novo Nordisk Investigational Site, Olten
  - Novo Nordisk Investigational Site, Schaffhausen
  - Novo Nordisk Investigational Site, Winterthur
  - Novo Nordisk Investigational Site, Zollikerberg
  - Novo Nordisk Investigational Site, Zurich

REFERENCES:
- [Result] Philis-Tsimikas A, Billings LK, Busch R, Portillo CM, Sahay R, Halladin N, Eggert S, Begtrup K, Harris S. Superior efficacy of insulin degludec/liraglutide versus insulin glargine U100 as add-on to sodium-glucose co-transporter-2 inhibitor therapy: A randomized clinical trial in people with uncontrolled type 2 diabetes. Diabetes Obes Metab. 2019 Jun;21(6):1399-1408. doi: 10.1111/dom.13666. Epub 2019 Apr 4. PMID 30761720
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 74 sites in 11 countries as follows: Argentina (3), Canada (5), Finland (6), Hungary (5), India (8), Russian Federation (7), Slovakia (5), Slovenia (4), Spain (6), Switzerland (5) and United States (20).
Pre-assignment Details: Subjects with type 2 diabetes mellitus on oral anti-diabetic drug (OAD) therapy with stable daily dose of sodium glucose co-transporter 2 inhibitors (SGLT2i) either as monotherapy or in combination with metformin ± dipeptidyl peptidase-4 inhibitors (DPP4i) ± pioglitazone according to locally approved label for at least 90 days prior to screening.
Groups:
- IDegLira: Subjects were administered with insulin degludec/liraglutide (IDegLira: 100 U/3.6 mg per mL) subcutaneously (s.c.) once daily for a duration of 26 weeks. IDegLira was supplied in a 3 mL prefilled PDS290 pen-injector with a fixed IDeg/liraglutide ratio of 100 U/3.6 mg per mL solution. IDegLira treatment was initiated at 10 dose steps (containing 10 units IDeg /0.36 mg liraglutide) and adjusted twice weekly on fixed days. Dose adjustment was based on the mean of three pre-breakfast self-measured plasma glucose (SMPG) values that were measured on the days of the titration and two days prior to the titration (target SMPG: 4.0-5.0 mmol/L [72 - 90 mg/dL]). The maximum daily dose was 50 dose steps (50 U IDeg /1.8 mg Lira). Pre-trial OAD treatments were continued according to current local label. The randomised subjects would be on either SGLT2i monotherapy or SGLT2i ± metformin ± pioglitazone, this treatment was to be unchanged throughout the trial, unless there was a safety concern.
- IGlar: Subjects were administered with insulin glargine (IGlar: 100 U/mL) subcutaneously (s.c.) once daily for a duration of 26 weeks. IGlar was supplied in a 3 mL pre-filled Solostar® pen at 100 U/mL solution. IGlar treatment was initiated with the starting dose of 10 U and adjusted twice weekly on fixed days. Dose adjustment was based on the mean of three pre-breakfast self-measured plasma glucose (SMPG) values measured on the days of the titration and two days prior to the titration (target SMPG: 4.0-5.0 mmol/L [72 - 90 mg/dL]). Pre-trial OAD treatments were continued according to current local label. The randomised subjects would be on either SGLT2i monotherapy or SGLT2i ± metformin ± pioglitazone, this treatment was to be unchanged throughout the trial, unless there was a safety concern.
Period: Overall Study
Arm/Group | IDegLira | IGlar
Started | 210 | 210
Exposed | 209 | 210
Completed | 200 | 206
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Unclassified | 1 | 1
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised".
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegLira | IGlar | Total
Number analyzed (Participants) | 210 | 210 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.4) | 57.2 (10.2) | 56.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 84 | 173
  Male | 121 | 126 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 37 | 68
  Not Hispanic or Latino | 179 | 173 | 352
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 31 | 35 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 175 | 171 | 346
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin)
Description: The mean change from baseline (week 0) in HbA1c values evaluated after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Number analysed = Number of subjects contributed to the analysis at baseline and week 26.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Percentage of glycosylated haemoglobin
  HbA1c (%) at baseline | 8.20 (0.93) | 8.36 (1.08)
  HbA1c (%) change from baseline to week 26: number analyzed (Participants) | 197 | 202
  HbA1c (%) change from baseline to week 26 | -1.94 (0.95) | -1.68 (1.05)
Statistical Analysis 1: Comparison: IDegLira vs IGlar; Analysis was based on ANCOVA model with treatment, pre-trial OAD, region as factors and baseline HbA1c as covariate. Data obtained after premature treatment discontinuation are included in the analysis. Missing data was imputed using unconditional reference based multiple imputation including data obtained after premature treatment discontinuation. The non-inferiority margin of 0.3 % was added to the end-of-treatment value for prematurely discontinued and withdrawn from trial IDegLira subjects; Test type: Non-Inferiority — Non-inferiority of IDegLira was considered confirmed if the upper limit of the two-sided 95% confidence interval (CI) for mean treatment difference (IDegLira minus IGlar) was strictly below 0.3%; ANCOVA; Treatment Contrast = -0.34, 95% CI 2-sided [-0.48 to -0.20] — IDegLira minus IGlar
Statistical Analysis 2: Comparison: IDegLira vs IGlar; This endpoint was analysed using an ANCOVA model with treatment, pre-trial OAD and region as factors and corresponding baseline value as covariate. Data obtained after premature treatment discontinuation were included in the analysis. Missing data were imputed using unconditional reference based multiple imputation including data obtained after premature treatment discontinuation; Test type: Superiority — Superiority of IDegLira was considered confirmed if the test procedure was not stopped (i.e. non-inferiority of IDegLira was confirmed for change from baseline in HbA1c; and superiority of IDegLira was confirmed for weight change and the number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes) and if the upper limit of the two-sided 95% CI for the mean treatment difference (IDegLira minus IGlar) in change from baseline in HbA1c was strictly below 0%; ANCOVA; Treatment Contrast = -0.36, 95% CI 2-sided [-0.50 to -0.21] — IDegLira minus IGlar

2. Secondary Outcome: Change in Body Weight
Description: The mean change from baseline (week 0) in body weight evaluated after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
kg
  Body weight (kg) at baseline | 89.3 (17.6) | 87.2 (17.2)
  Body weight (kg) change from baseline to week 26: number analyzed (Participants) | 199 | 204
  Body weight (kg) change from baseline to week 26 | -0.0 (3.8) | 2.0 (3.9)
Statistical Analysis 1: Comparison: IDegLira vs IGlar; This endpoint was analysed using an ANCOVA model with treatment, pre-trial OAD and region as factors and corresponding baseline weight as covariate. Data obtained after premature treatment discontinuation were included in the analysis. Missing data were imputed using unconditional reference based multiple imputation including data obtained after premature treatment discontinuation; Test type: Superiority — Superiority of IDegLira was considered confirmed if the test procedure was not stopped (i.e. non-inferiority of IDegLira was confirmed for change from baseline in HbA1c) and if the upper limit of the two-sided 95% CI for the mean treatment difference (IDegLira minus IGlar) in change from baseline in body weight was strictly below 0 kg; ANCOVA; Treatment Contrast = -1.92, 95% CI 2-sided [-2.64 to -1.19] — IDegLira minus IGlar

3. Secondary Outcome: Number of Treatment-emergent Severe or BG (Blood Glucose) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe (subjects who were not able to self-treat) and/or BG confirmed by a plasma glucose values <3.1 mmol/L (56 mg/dL) with accompanied symptoms consistent with hypoglycaemia.
Time Frame: Week 0-26
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of episodes | 38 | 95
Statistical Analysis 1: Comparison: IDegLira vs IGlar; This endpoint was analysed using a negative binomial regression model with a log link and the logarithm of the exposure time as offset. The model included treatment and pre-trial OAD as fixed factors. Missing data were imputed using multiple imputations (conditioning on expected event rate before premature treatment discontinuation or withdrawal from trial as if treated with IGlar); Test type: Superiority — Superiority of IDegLira was considered confirmed if the test procedure was not stopped (i.e. non-inferiority of IDegLira was confirmed for change from baseline in HbA1c and superiority of IDegLira was confirmed for change from baseline in body weight) and if the upper limit of the two-sided 95% CI for the rate ratio (IDegLira over IGlar) of rate of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes was strictly below 1; Negative binomial regression model; Treatment Ratio = 0.42, 95% CI 2-sided [0.23 to 0.75] — IDegLira over IGlar

4. Secondary Outcome: Insulin Dose, Total Daily Dose (U)
Description: Actual daily total insulin dose (Units) was evaluated after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Number analysed = Number of subjects contributed to the analysis at week 26.
Measure: Mean (Standard Deviation); unit: Units (U)
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Units (U) | 36.2 (13.4) | 53.5 (26.1)
Statistical Analysis 1: Comparison: IDegLira vs IGlar; The endpoint was analysed using an ANCOVA model with treatment, pre-trial OAD and region as factors and corresponding baseline HbA1c as covariate. Missing data were imputed using unconditional reference based multiple imputation including data obtained after premature treatment discontinuation; Test type: Superiority — Superiority of IDegLira was considered confirmed if the test procedure was not stopped (i.e. non-inferiority of IDegLira was confirmed for change from baseline in HbA1c; and superiority of IDegLira was confirmed for weight change, number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes and change in HbA1c) and if the upper limit of the two-sided 95% CI for the mean treatment difference (IDegLira minus IGlar) in insulin dose after 26 weeks was strictly below 0 U; ANCOVA; Treatment Contrast = -15.37, 95% CI 2-sided [-19.60 to -11.13] — IDegLira minus IGlar

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG was evaluated after 26 weeks of randomised treatment.
Time Frame: Week 0, Week 26
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Number analysed = Number of subjects contributed to the analysis at baseline (week 0) and week 26.
Measure: Mean (Standard Deviation); unit: mmol/ L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/ L
  FPG (mmol/L) at baseline: number analyzed (Participants) | 206 | 206
  FPG (mmol/L) at baseline | 9.51 (2.69) | 9.57 (2.40)
  FPG (mmol/L) change from baseline to week 26: number analyzed (Participants) | 189 | 195
  FPG (mmol/L) change from baseline to week 26 | -3.72 (2.89) | -3.50 (2.43)

6. Secondary Outcome: Number of Treatment-emergent Adverse Events
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 26. TEAE was defined as an event that has onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Week 0-26
Population: as for outcome 3
Measure: Number; unit: Number of events
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of events | 450 | 386

7. Secondary Outcome: Responder (Yes/No) for HbA1c Below 7.0%
Description: The proportion of subjects achieving pre-defined HbA1c targets <7.0% after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 167 | 144
  No: number analyzed (Participants) | 197 | 202
  No | 30 | 58

8. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c < 7.0% Without Weight Gain
Description: The proportion of subjects achieving pre-defined HbA1c targets <7.0% without weight gain after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 91 | 38
  No: number analyzed (Participants) | 197 | 202
  No | 106 | 164

9. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c < 7.0% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: The proportion of subjects achieving pre-defined HbA1c targets <7.0% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 156 | 114
  No: number analyzed (Participants) | 197 | 202
  No | 41 | 88

10. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c < 7.0% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment and Without Weight Gain
Description: The proportion of subjects achieving pre-defined HbA1c targets <7.0% without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment and without weight gain. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 83 | 34
  No: number analyzed (Participants) | 197 | 202
  No | 114 | 168

11. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c ≤ 6.5%
Description: The proportion of subjects achieving pre-defined HbA1c targets ≤ 6.5% after 26 weeks of randomised treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 147 | 100
  No: number analyzed (Participants) | 197 | 202
  No | 50 | 102

12. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c ≤ 6.5% Without Weight Gain
Description: The proportion of subjects achieving pre-defined HbA1c targets ≤ 6.5% without weight gain after 26 weeks of randomised treatment. The results are based on retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Participants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 84 | 26
  No: number analyzed (Participants) | 197 | 202
  No | 113 | 176

13. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c ≤ 6.5% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: The proportion of subjects achieving pre-defined HbA1c targets ≤ 6.5%without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Particpants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Particpants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 137 | 79
  No: number analyzed (Participants) | 197 | 202
  No | 60 | 123

14. Secondary Outcome: Responder After 26 Weeks (Yes/No) for: HbA1c ≤ 6.5% Without Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment and Without Weight Gain
Description: The proportion of subjects achieving pre-defined HbA1c targets ≤ 6.5%without treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment and without weight gain. The results presented included retrieved data at week 26 for subjects who prematurely discontinued the trial product.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Number; unit: Partcipants
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Partcipants
  Yes: number analyzed (Participants) | 197 | 202
  Yes | 77 | 24
  No: number analyzed (Participants) | 197 | 202
  No | 120 | 178

15. Secondary Outcome: Change From Baseline After 26 Weeks in Waist Circumference
Description: Mean change from baseline in waist circumference after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
cm
  Waist circum. (cm) at baseline | 105.9 (12.7) | 104.7 (11.3)
  Waist circum. (cm) change from baseline to week 26: number analyzed (Participants) | 194 | 200
  Waist circum. (cm) change from baseline to week 26 | -0.6 (4.6) | 0.7 (3.9)

16. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Cholesterol
Description: The values of total cholesterol from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 4
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Total cholesterol (mmol/L) at baseline: number analyzed (Participants) | 206 | 205
  Total cholesterol (mmol/L) at baseline | 4.42 [2.02 to 10.62] | 4.45 [2.12 to 11.37]
  Total cholesterol (mmol/L) at week 26: number analyzed (Participants) | 191 | 199
  Total cholesterol (mmol/L) at week 26 | 4.27 [2.12 to 9.87] | 4.27 [1.84 to 9.40]

17. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Low-density Lipoprotein Cholesterol (LDL Cholesterol)
Description: The values of LDL cholesterol from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  LDL cholesterol (mmol/L) at baseline: number analyzed (Participants) | 205 | 205
  LDL cholesterol (mmol/L) at baseline | 2.28 [0.26 to 7.10] | 2.28 [0.10 to 6.73]
  LDL cholesterol (mmol/L) at week 26: number analyzed (Participants) | 191 | 199
  LDL cholesterol (mmol/L) at week 26 | 2.20 [0.57 to 6.42] | 2.31 [0.62 to 5.34]

18. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: High-density Lipoprotein Cholesterol (HDL Cholesterol)
Description: The values of HDL cholesterol from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  HDL cholesterol (mmol/L) at baseline: number analyzed (Participants) | 206 | 205
  HDL cholesterol (mmol/L) at baseline | 1.14 [0.57 to 2.69] | 1.14 [0.31 to 2.59]
  HDL cholesterol (mmol/L) at week 26: number analyzed (Participants) | 191 | 199
  HDL cholesterol (mmol/L) at week 26 | 1.17 [0.57 to 2.72] | 1.17 [0.36 to 2.49]

19. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Very-low-density Lipoprotein Cholesterol (VLDL Cholesterol)
Description: The values of VLDL cholesterol from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  VLDL cholesterol (mmol/L) at baseline: number analyzed (Participants) | 205 | 205
  VLDL cholesterol (mmol/L) at baseline | 0.75 [0.18 to 8.60] | 0.80 [0.21 to 8.13]
  VLDL cholesterol (mmol/L) at week 26: number analyzed (Participants) | 191 | 199
  VLDL cholesterol (mmol/L) at week 26 | 0.70 [0.21 to 5.75] | 0.67 [0.21 to 3.32]

20. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Triglycerides
Description: The values of triglycerides from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Triglycerides (mmol/L) at baseline: number analyzed (Participants) | 206 | 205
  Triglycerides (mmol/L) at baseline | 1.67 [0.38 to 23.60] | 1.73 [0.43 to 27.80]
  Triglycerides (mmol/L) at week 26: number analyzed (Participants) | 191 | 199
  Triglycerides (mmol/L) at week 26 | 1.55 [0.46 to 17.03] | 1.47 [0.47 to 8.81]

21. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Free Fatty Acids
Description: The values of free fatty acids from fasting lipid profile after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Free fatty acids (mmol/L) at baseline: number analyzed (Participants) | 204 | 207
  Free fatty acids (mmol/L) at baseline | 0.58 [0.08 to 1.44] | 0.61 [0.06 to 1.73]
  Free fatty acids (mmol/L) at week 26: number analyzed (Participants) | 189 | 199
  Free fatty acids (mmol/L) at week 26 | 0.38 [0.10 to 0.92] | 0.42 [0.02 to 1.30]

22. Secondary Outcome: Change From Baseline in the 9-point Self-measured Plasma Glucose (SMPG) Profile
Description: Change in 9-point SMPG profile was evaluated after 26 weeks of randomised treatment. SMPG measurements at baseline and week 26 are presented here at the following mentioned time points:1) Before breakfast, 2) 90 mins after the start of Breakfast, 3) Before lunch, 4) 90 mins after the start of lunch, 5) Before dinner, 6) 90 mins after the start of dinner, 7) At bedtime, 8) At 4 AM, 9) Before breakfast the following day.
Time Frame: After 26 weeks
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Number analysed = Number of subjects contributed to the analysis at baseline and week 26 for mentioned time points.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Before breakfast - Baseline: number analyzed (Participants) | 210 | 207
  Before breakfast - Baseline | 9.01 (2.18) | 9.00 (1.91)
  Ninety (90) minutes after breakfast - Baseline: number analyzed (Participants) | 209 | 207
  Ninety (90) minutes after breakfast - Baseline | 11.79 (3.09) | 11.77 (2.99)
  Before lunch - Baseline: number analyzed (Participants) | 208 | 207
  Before lunch - Baseline | 8.93 (2.80) | 9.20 (2.95)
  Ninety (90) minutes after lunch - Baseline: number analyzed (Participants) | 210 | 207
  Ninety (90) minutes after lunch - Baseline | 11.24 (3.26) | 11.22 (3.06)
  Before dinner - Baseline: number analyzed (Participants) | 210 | 206
  Before dinner - Baseline | 9.33 (2.70) | 9.36 (2.89)
  Ninety (90) minutes after dinner - Baseline: number analyzed (Participants) | 205 | 206
  Ninety (90) minutes after dinner - Baseline | 11.40 (3.04) | 11.40 (2.99)
  At bedtime - Baseline: number analyzed (Participants) | 202 | 202
  At bedtime - Baseline | 10.38 (3.16) | 10.71 (3.13)
  At 4.00 AM - Baseline: number analyzed (Participants) | 198 | 201
  At 4.00 AM - Baseline | 8.80 (2.41) | 9.00 (2.50)
  Before breakfast the following day - Baseline: number analyzed (Participants) | 204 | 207
  Before breakfast the following day - Baseline | 8.60 (2.02) | 8.81 (1.92)
  Before breakfast - Week 26: number analyzed (Participants) | 184 | 188
  Before breakfast - Week 26 | 5.40 (1.24) | 5.39 (1.21)
  Ninety (90) minutes after breakfast - Week 26: number analyzed (Participants) | 182 | 187
  Ninety (90) minutes after breakfast - Week 26 | 7.20 (1.86) | 8.35 (2.40)
  Before lunch - Week 26: number analyzed (Participants) | 182 | 187
  Before lunch - Week 26 | 5.83 (1.36) | 6.35 (1.88)
  Ninety (90) minutes after lunch - Week 26: number analyzed (Participants) | 179 | 187
  Ninety (90) minutes after lunch - Week 26 | 7.25 (1.73) | 8.49 (2.28)
  Before dinner - Week 26:: number analyzed (Participants) | 181 | 186
  Before dinner - Week 26: | 6.43 (1.61) | 6.77 (2.03)
  Ninety (90) minutes after dinner - Week 26: number analyzed (Participants) | 180 | 186
  Ninety (90) minutes after dinner - Week 26 | 7.85 (1.95) | 8.70 (2.19)
  At bedtime - Week 26: number analyzed (Participants) | 173 | 183
  At bedtime - Week 26 | 7.05 (1.91) | 7.79 (2.20)
  At 4.00 AM - Week 26: number analyzed (Participants) | 175 | 178
  At 4.00 AM - Week 26 | 5.58 (1.17) | 5.72 (1.51)
  Before breakfast the following day - Week 26: number analyzed (Participants) | 180 | 188
  Before breakfast the following day - Week 26 | 5.23 (1.09) | 5.36 (1.38)

23. Secondary Outcome: Change From Baseline in Self-measured Plasma Glucose (SMPG) 9-point Profile: Mean of the 9-point Profile
Description: Change in mean of the 9-point profile SMPG was evaluated after 26 weeks of randomised treatment. 9-point profile SMPG was measured at the following mentioned time points:1) Before breakfast, 2) 90 mins after the start of Breakfast, 3) Before lunch, 4) 90 mins after the start of lunch, 5) Before dinner, 6) 90 mins after the start of dinner, 7) At bedtime, 8) At 4 AM, 9) Before breakfast the following day.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Mean 9-point SMPG (mmol/L) at baseline: number analyzed (Participants) | 204 | 207
  Mean 9-point SMPG (mmol/L) at baseline | 9.98 (2.17) | 10.06 (2.04)
  Mean 9-point SMPG change from baseline to week 26: number analyzed (Participants) | 176 | 185
  Mean 9-point SMPG change from baseline to week 26 | -3.47 (2.01) | -2.98 (1.91)

24. Secondary Outcome: Change From Baseline in SMPG 9-point Profile: Prandial Plasma Glucose Increments (From Before Meal to 90 Min After Breakfast, Lunch and Dinner). The Mean Increment Over All Meals Will be Derived as the Mean of All Available Meal Increments
Description: Mean prandial plasma glucose increments for each meal (from before meal to 90 min after breakfast, lunch and dinner) was evaluated after 26 weeks of randomised treatment. The mean increment over all meals was derived as the mean of all available meal increments are presented here.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmol/L
  Baseline: number analyzed (Participants) | 210 | 207
  Baseline | 2.38 (1.73) | 2.28 (1.88)
  Change from baseline to week 26: number analyzed (Participants) | 182 | 185
  Change from baseline to week 26 | -0.86 (1.95) | -0.09 (1.96)

25. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from baseline (week 0) in systolic blood pressure (BP) was evaluated after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmHg
  Systolic BP (mmHg) at baseline | 130.5 (14.3) | 128.9 (13.1)
  Systolic BP (mmHg) change from baseline to week 26: number analyzed (Participants) | 194 | 200
  Systolic BP (mmHg) change from baseline to week 26 | -3.0 (12.7) | 0.6 (12.0)

26. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from baseline (week 0) in diastolic blood pressure was evaluated after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
mmHg
  Diastolic (mmHg) at baseline | 79.4 (8.0) | 78.9 (8.9)
  Diastolic (mmHg) change from baseline to week 26: number analyzed (Participants) | 194 | 200
  Diastolic (mmHg) change from baseline to week 26 | -1.2 (8.4) | -1.1 (8.3)

27. Secondary Outcome: Number of Treatment-emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During 26 Weeks
Description: Number of treatment-emergent nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes (00:01-05:59 - inclusive) during 26 weeks of randomised treatment.
Time Frame: Week 0-26
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of episodes | 6 | 13

28. Secondary Outcome: Number of Treatment-emergent Hypoglycaemic Episodes According to ADA Definition During 26 Weeks
Description: American Diabetes Association (ADA) classification of hypoglycaemic episodes: 1)Severe: Requiring assistance of another person to actively administer carbohydrate/glucagon/take other corrective actions. PG levels may not be available during an event, but neurological recovery following return of PG to normal is considered sufficient evidence that event was induced by a low PG level. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo: PG >3.9 mmol/L with symptoms. 6) Unclassifiable.
Time Frame: Week 0-26
Population: as for outcome 27
Measure: Number; unit: Number of episodes
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of episodes
  Severe - ADA | 1 | 0
  Documented symptomatic - ADA | 239 | 419
  Asymptomatic - ADA | 850 | 902
  Probably symptomatic - ADA | 23 | 5
  Pseudo - ADA | 10 | 14
  Unclassifiable hypoglycaemia - ADA | 2 | 0

29. Secondary Outcome: Change From Baseline in Clinical Evaluation After 26 Weeks: Electrocardiogram (ECG)
Description: Reported results are ECG findings at screening and week 26 of randomised treatment. Since the values measured at the baseline (week 0) were not collected, the screening data (week -2, which is <= 2 weeks before baseline) is presented here. The findings are categorised as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). 4) Missing.
Time Frame: After 26 weeks
Population: The safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated". Number analysed = Number of subjects contributed to the analysis at screening and week 26.
Measure: Number; unit: Number of subjects
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of subjects
  Screening, Normal | 142 | 141
  Screening, Abnormal NCS | 66 | 69
  Screening, Abnormal CS | 1 | 0
  Screening, Missing | 0 | 0
  Week 26, Normal: number analyzed (Participants) | 194 | 200
  Week 26, Normal | 134 | 136
  Week 26, Abnormal NCS: number analyzed (Participants) | 194 | 200
  Week 26, Abnormal NCS | 58 | 64
  Week 26, Abnormal CS: number analyzed (Participants) | 194 | 200
  Week 26, Abnormal CS | 2 | 0
  Week 26, Missing: number analyzed (Participants) | 194 | 200
  Week 26, Missing | 0 | 0

30. Secondary Outcome: Change From Baseline in Clinical Evaluation After 26 Weeks: Eye Examination: Fundoscopy/Fundus Photography
Description: Reported results are fundus photography/fundoscopy (for both left and right eye) findings at screening and week 26 of randomised treatment. Since the values measured at the baseline (week 0) were not collected, the screening data (week -2, which is <= 2 weeks before baseline) is presented here. The findings are categorised as: 1) Normal. 2) Abnormal (not clinically significant [NCS]). 3) Abnormal (clinically significant [CS]). 4) Missing.
Time Frame: After 26 weeks
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated". Number analysed = Number of subjects contributed to the analysis at screening and week 26.
Measure: Number; unit: Number of subjects
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Number of subjects
  Screening, Left eye (Normal): number analyzed (Participants) | 209 | 209
  Screening, Left eye (Normal) | 134 | 131
  Screening, Left eye (Abnormal -NCS): number analyzed (Participants) | 209 | 209
  Screening, Left eye (Abnormal -NCS) | 68 | 74
  Screening, Left eye (Abnormal-CS): number analyzed (Participants) | 209 | 209
  Screening, Left eye (Abnormal-CS) | 7 | 4
  Screening, Left eye (Missing): number analyzed (Participants) | 209 | 209
  Screening, Left eye (Missing) | 0 | 0
  Week 26, Left eye (Normal): number analyzed (Participants) | 191 | 197
  Week 26, Left eye (Normal) | 123 | 125
  Week 26, Left eye (Abnormal -NCS): number analyzed (Participants) | 191 | 197
  Week 26, Left eye (Abnormal -NCS) | 66 | 68
  Week 26, Left eye (Abnormal-CS): number analyzed (Participants) | 191 | 197
  Week 26, Left eye (Abnormal-CS) | 2 | 4
  Week 26, Left eye (Missing): number analyzed (Participants) | 191 | 197
  Week 26, Left eye (Missing) | 0 | 0
  Screening, Right eye (Normal): number analyzed (Participants) | 209 | 209
  Screening, Right eye (Normal) | 133 | 133
  Screening, Right eye (Abnormal-NCS): number analyzed (Participants) | 209 | 209
  Screening, Right eye (Abnormal-NCS) | 69 | 72
  Screening, Right eye (Abnormal- CS): number analyzed (Participants) | 209 | 209
  Screening, Right eye (Abnormal- CS) | 7 | 4
  Screening, Right eye (Missing): number analyzed (Participants) | 209 | 209
  Screening, Right eye (Missing) | 0 | 0
  Week 26, Right eye (Normal): number analyzed (Participants) | 191 | 197
  Week 26, Right eye (Normal) | 120 | 127
  Week 26, Right eye (Abnormal-NCS): number analyzed (Participants) | 191 | 197
  Week 26, Right eye (Abnormal-NCS) | 69 | 66
  Week 26, Right eye (Abnormal- CS): number analyzed (Participants) | 191 | 197
  Week 26, Right eye (Abnormal- CS) | 2 | 4
  Week 26, Right eye (Missing): number analyzed (Participants) | 191 | 197
  Week 26, Right eye (Missing) | 0 | 0

31. Secondary Outcome: Change From Baseline in Clinical Evaluation After 26 Weeks: Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated after 26 weeks of randomised treatment.
Time Frame: After 26 weeks
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or comparator. Subjects in the safety set contributed to the evaluation "as treated". Number analysed = Number of subjects contributed to the analysis at baseline (week 0) and week 26.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 209 | 210
Beats/minute
  Pulse (beats/min) at baseline | 76.1 (9.1) | 75.0 (9.5)
  Pulse (beats/min) change from baseline to week 26: number analyzed (Participants) | 194 | 200
  Pulse (beats/min) change from baseline to week 26 | 2.0 (8.4) | -0.4 (8.2)

32. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) After 26 Weeks: Summary Scores of Medical Outcomes Study 36-item Short Form (SF-36v2)
Description: The Short Form (SF)-36v2™ patient reported outcomes (PRO) questionnaire was used to assess the subject's overall health related quality of life (HRQoL). PRO questionnaire (SF-36v2™) measured the HRQoL which contains 36 items covering 8 domains of physical and mental health status. The raw scale scores from the SF-36 were transformed to a 0-100 scale scores (where higher scores indicated a better health status) which is further converted to norm-based scores using a T-score transformation in order to obtain a direct interpretation in relation to the distribution of the scores in the 2009 reference population . The total/overall (SF-36v2™) scores for physical and mental health from baseline to week 26 are presented here.
Time Frame: After 26 weeks
Population: The FAS included all randomised subjects. The statistical evaluation of the FAS followed the intent-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Number analysed = Number of subjects contributed to the analysis at baseline and week 26 for overall physical and mental scores.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Scores on a scale
  Overall physical - Baseline: number analyzed (Participants) | 208 | 209
  Overall physical - Baseline | 51.3 [22.0 to 61.6] | 51.5 [21.9 to 62.4]
  Overall physical - Week 26: number analyzed (Participants) | 194 | 200
  Overall physical - Week 26 | 53.2 [22.9 to 64.0] | 54.6 [25.0 to 65.6]
  Overall mental - Baseline: number analyzed (Participants) | 208 | 210
  Overall mental - Baseline | 53.3 [15.6 to 67.9] | 53.3 [19.7 to 68.8]
  Overall mental - Week 26: number analyzed (Participants) | 194 | 200
  Overall mental - Week 26 | 54.4 [14.8 to 68.3] | 54.4 [31.0 to 67.3]

33. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) After 26 Weeks: Summary Scores of Treatment Related Impact Measure for Diabetes (TRIM-D)
Description: The patient reported outcomes are calculated based on TRIM-D questionnaire. The TRIM-D questionnaire consists of 5 sub-domains (treatment burden, daily life, diabetes management, compliance and psychological health), where each question is scored to a 1-5-point scale with a higher score indicating a better health state (less negative impact). Mean TRIM-D domain scores and the total scores are later transformed to a 0-100 scale for analysis. Summary scores from baseline and week 26 for total/overall scores are presented here.
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | IDegLira | IGlar
Number analyzed (Participants) | 210 | 210
Scores on a scale
  TRIM-D scores at baseline: number analyzed (Participants) | 208 | 210
  TRIM-D scores at baseline | 75.9 [44.6 to 100.0] | 75.9 [38.4 to 100.0]
  TRIM-D scores at week 26: number analyzed (Participants) | 194 | 199
  TRIM-D scores at week 26 | 84.4 [37.5 to 100.0] | 83.9 [44.6 to 100.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first day (week 0) of exposure to randomised treatment of 26 weeks + 30 days follow-up visits after the last dose on trial product. All reported AEs are treatment emergent (i.e., TEAE).
Description: Results are based on the safety analysis set, which included all subjects who received at least one dose of the investigational product or its comparator. Subjects in the safety set contributed to the evaluation "as treated".
Arm/Group | IDegLira | IGlar
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/210
Serious Adverse Events (participants affected / at risk) | 6/209 | 7/210
Other Adverse Events (participants affected / at risk) | 49/209 | 45/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=209) | IGlar (N=210)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular evaluation (Investigations) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Device failure (Product Issues) | 1 (2) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=209) | IGlar (N=210)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (15)
Headache (Nervous system disorders) | 18 (35) | 19 (27)
Lipase increased (Investigations) | 12 (15) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (22) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 16 (22) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property".

DOCUMENTS (2):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02773368/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02773368/SAP_001.pdf